CLINICAL TRIAL: NCT03899545
Title: Does Serratus Plane Plus Pectoral I Block Provide Better Perioperative Analgesia in Ambulatory Breast Cancer Surgery When Compared to Serratus Plane Block Alone
Brief Title: Serratus Plane Plus Pectoral I Block Versus Serratus Plane Block for Perioperative Analgesia in Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Serdar Yeşiltaş, Lecturer, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 71306642-5/24
Record Dates: First submitted 2019-03-31; First posted 2019-04-02 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain; Postoperative Nausea; Patient Satisfaction; Narcotic Use
Keywords: serratus plane block; pectoral I block; breast cancer surgery; perioperative analgesia
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Serratus Plane Block (Experimental): Serratus plane block will be applied after induction of general anesthesia.
  Interventions: Other: Serratus Plane Block
- Serratus Plane Block plus Pectoral I block (Active Comparator): Serratus plane plus pectoral I block will be applied after induction of general anesthesia.
  Interventions: Other: Serratus Plane Block plus Pectoral I Block

INTERVENTIONS:
Other: Serratus Plane Block — 0.5 ml /kg Bupivacaine/lidocaine mixture will be injected onto the serratus muscle
  Arms: Serratus Plane Block
Other: Serratus Plane Block plus Pectoral I Block — 0.5 ml / kg %0.25 Bupivacaine/ %1 lidocaine mixture will be injected onto the serratus muscle and injected between the pectoralis minor/pectoralis major muscles.2/3 of the total drug will be applied for the serratus plane block and 1/3 of the total drug for the pectoral I block. If the total amount of the drug is less than 30 ml, it will be completed with isotonic saline to 30 ml.
  Arms: Serratus Plane Block plus Pectoral I block

SUMMARY:
Breast cancer is the most common malignancy in women at worldwide. Even a minor breast surgery can cause significant postoperative pain (PP) (1). PP could be converted into chronic pain in 25-40% of cases. Inadequate PP control is associated with increased morbidity, delay in wound healing, prolonged hospital stay, increased opioid use, increased side effects and high cost of care. For these reasons, regional anesthetic techniques are recommended for effective PP management. Some of recent studies suggest that ultrasound-guided pectoral I (PI), pectoral II (PII) and serratus plan block (SPB) may be an alternative to thoracic epidural analgesia and paravertebral block applications because of the ease of administration, low side effect profile and adequate analgesia in breast surgery. (2,3).

DETAILED DESCRIPTION:
In breast surgeries, the serratus plane block has recently been described and rapidly became popular. The serratus plane block is called the modified pectoral II block. Local anesthetic drugs are injected onto the serratus muscle by targeting thoracodorsal nerve, thoracicus longus nerve, lateral and anterior branches of the T2-T9 intercostal nerves. In the pectoral I (Pecs I) block, the medial and lateral pectoral nerves of the brachial plexus are targeted. Additionally, Pecs I block can be effective for analgesia in axillary dissection. In the literature, there are studies comparing pectoral I + II blocks and serratus plane block in terms of analgesic efficacy in breast surgery. The aim of this study was to evaluate the postoperative analgesic efficiency of serratus plane block and serratus plan block plus pectoral I block combination.

Participans will be informed about the potential benefits and complications after the study protocol has been fully and thoroughly explained. After premedication with 0.03 mg / kg iv midazolam, participans will be noninvasively monitored by taking into the operating room (heart rate, blood pressure, pulse oximetry). Anesthesia induction will delivered with fentanyl 1mcg / kg, propofol 1.5-2 mg / kg and rocuronium 0.5 mg / kg. The maintenance of anesthesia will be achieved by infusion of sevoflurane 1-3% in 50% O2/50% medical air. The depth of anesthesia will be evaluated with bispectral index monitoring and will be kept between 40 and 60.. Thirty minutes before end of the surgery, all patients were intravenously administered 20 mg tenoxicam HCl and 1gr paracetamol.

SPB plus Pecs I block technique: Bupivacaine/lidocaine mixture will be injected onto the serratus muscle and injected between the pectoralis minor/pectoralis major muscles.

SPB technique: Bupivacaine/lidocaine mixture will be injected onto the serratus muscle.

After the surgery, 1 g paracetamol was intravenously administered once every 8 h. Postoperative pain was assessed using VAS (VAS 0 = no pain, VAS 10 = most severe pain ). Morphine 0.1mg / kg will be used as rescue analgesic drug.Duration at PACU was recorded right from 0 h. VAS scores at 0, 1,2, 6, 12 and 24 h were recorded. PONV was evaluated using a numeric ranking scale (0 = no PONV, 1 = mild nausea, 2 = severe nausea or vomiting once attack, and 3 = vomiting more than once attack). If PONV score was >2, the antiemetic metoclopramide Hcl 10mg was intravenously administered.

ELIGIBILITY:
Inclusion Criteria:

1. ASA 1-2-3
2. Patients scheduled for elective surgery

Exclusion Criteria:

1. Previous neurological disease symptom (TIA, syncope, dementia, etc.)
2. Allergy to drugs
3. Major cardiac disease
4. Renal failure
5. Psychiatric disease
6. Patients who refuse to participate in the study

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-06 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Pain intensity score | 24 hour
  Self reported pain intensity in the postoperative 0, 1,2,6,12 and 24 hour. Each item is scored 0-10 (0: no pain 10: pain as bad as can be)

SECONDARY OUTCOMES:
İntraoperative fentanyl requirement | during surgery
  Total amount of fentanyl use
time to first analgesic request | 24 hour
  time to first analgesic use
Postoperative opioid consumption | 24 hour
  If pain intensity score >4 morphine 0,1 mg/kg will be given to the patient. The total amount of morphine requirement will be recorded.
Postoperative nausea and vomiting | 24 hour
  Nausea and vomiting intensity score measured by numeric rank score (0:no nausea and no vomiting, 1: have nausea, no vomiting, 2: once vomiting, 3: two or more vomiting).
Patient satisfaction: score | 24 hour
  Will be scored between 1-5 (1- very bad 5-very good).

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Yeşiltaş, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yesiltas S, Turkoz A, Calim M, Yilmaz S, Esen A, Daskaya H, Karaaslan K. Comparison of serratus plane block alone and in combination with pectoral type 1 block for breast cancer surgery: a randomized controlled study. Hippokratia. 2021 Jan-Mar;25(1):8-14. PMID 35221650